CLINICAL TRIAL: NCT02412761
Title: Series of N-of-1 Crossover Trials of Antihypertensive Therapy in Adolescents With Essential Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Joyce Philip Samuel, Assistant Professor of Pediatrics, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-13-0287; 5KL2TR000370 (NIH)
Record Dates: First submitted 2015-04-03; First posted 2015-04-09 (Estimated); Results first posted 2018-11-15 (Actual); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Essential Hypertension
Keywords: Anti-hypertensive medications; Pediatrics; N-of-1 trial
MeSH Terms: conditions — Essential Hypertension | interventions — Lisinopril; Angiotensin-Converting Enzyme Inhibitors; Amlodipine; Hydrochlorothiazide; Sodium Chloride Symporter Inhibitors

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (6):
- Amlodipine, then HCTZ, then Lisinopril (Active Comparator): Participants first received amlodipine once daily for 2 weeks, then crossed over to hydrochlorothiazide (HCTZ) once daily for 2 weeks, then lisinopril once daily for 2 weeks. Subsequent treatments varied depending on individual patient response.
  Interventions: Drug: Lisinopril; Drug: Amlodipine; Drug: Hydrochlorothiazide
- Amlodipine, then Lisinopril, then HCTZ (Active Comparator): Participants first received amlodipine once daily for 2 weeks, then crossed over to lisinopril once daily for 2 weeks, then hydrochlorothiazide (HCTZ) once daily for 2 weeks. Subsequent treatments varied depending on individual patient response.
  Interventions: Drug: Lisinopril; Drug: Amlodipine; Drug: Hydrochlorothiazide
- HCTZ, then Amlodipine, then Lisinopril (Active Comparator): Participants first received hydrochlorothiazide (HCTZ) once daily for 2 weeks, then crossed over to amlodipine once daily for 2 weeks, then lisinopril once daily for 2 weeks. Subsequent treatments varied depending on individual patient response.
  Interventions: Drug: Lisinopril; Drug: Amlodipine; Drug: Hydrochlorothiazide
- HCTZ, then Lisinopril, then Amlodipine (Active Comparator): Participants first received hydrochlorothiazide (HCTZ) once daily for 2 weeks, then crossed over to lisinopril once daily for 2 weeks, then amlodipine once daily for 2 weeks. Subsequent treatments varied depending on individual patient response.
  Interventions: Drug: Lisinopril; Drug: Amlodipine; Drug: Hydrochlorothiazide
- Lisinopril, then Amlodipine, then HCTZ (Active Comparator): Participants first received lisinopril once daily for 2 weeks, then crossed over to amlodipine once daily for 2 weeks, then hydrochlorothiazide (HCTZ) once daily for 2 weeks. Subsequent treatments varied depending on individual patient response.
  Interventions: Drug: Lisinopril; Drug: Amlodipine; Drug: Hydrochlorothiazide
- Lisinopril, then HCTZ, then Amlodipine (Active Comparator): Participants first received lisinopril once daily for 2 weeks, then crossed over to hydrochlorothiazide (HCTZ) once daily for 2 weeks, then amlodipine once daily for 2 weeks. Subsequent treatments varied depending on individual patient response.
  Interventions: Drug: Lisinopril; Drug: Amlodipine; Drug: Hydrochlorothiazide

INTERVENTIONS:
Drug: Lisinopril — Initial dose: 0.1 mg/kg/dose orally, once daily (maximum initial dose 10 mg/dose). Maximum final dose: 40 mg/dose or 0.6 mg/kg/dose.
  Other Names: Angiotensin-converting enzyme inhibitor
Drug: Amlodipine — Initial dose: 0.1 mg/kg/dose orally, once daily (maximum initial dose 5 mg/dose). Maximum final dose: 10 mg/dose
  Other Names: Dihydropyridine calcium channel blocker
Drug: Hydrochlorothiazide — Initial dose: 1 mg/kg/dose orally, once daily (maximum initial dose 25 mg/dose). Maximum final dose: 50 mg/dose or 3 mg/kg/dose
  Other Names: Thiazide diuretic

SUMMARY:
Children are increasingly being diagnosed with essential hypertension and the absence of comparative effectiveness research in antihypertensive therapies has contributed to considerable differences in prescribing practices among physicians treating children with essential hypertension.

This study will consist of a series of systematically-administered n-of-1 trials among children to verify the need for ongoing antihypertensive treatment and if so, to identify the preferred single drug therapy.

DETAILED DESCRIPTION:
This is a series of systematically-administered n-of-1 trials among children with essential hypertension to verify the need for ongoing antihypertensive treatment and if so, to identify the preferred single drug therapy from among the three major classes of drugs commonly used for essential hypertension (angiotensin converting enzyme inhibitors, calcium channel blockers, and diuretics). The investigators will determine whether there is one that is preferred for the great majority of patients. The "preferred" therapy will be defined as the drug which produces normal ambulatory blood pressure, with the greatest reduction in awake mean systolic blood pressure without unacceptable side effects.

For each patient, the order of the 3 drugs will be assigned randomly and each drug will be taken for 2 weeks. The effectiveness of each drug will be measured with 24-hour ambulatory blood pressure monitoring, and tolerability will be assessed using a side effect questionnaire. Participants will rotate through treatment periods, repeating drugs and adjusting doses until the preferred therapy is identified. In assessing whether one the medications is most effective for the great majority of subjects, the primary outcome will be the percentage of participants for whom each drug is selected as the preferred therapy. Primary hypothesis: no drug will be selected for the majority of the subjects, a finding that would support consideration of clinical use of n-of-1 trials. Secondary analyses will explore whether patient characteristics predict which medication will be selected as a preferred drug.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of essential hypertension
* Treating physician has determined that pharmacologic therapy is necessary

Exclusion Criteria:

* Compelling indication to select one particular medication
* Specific contraindication for any of the 3 therapies

Ages: 9 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2013-06; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joyce P Samuel, MD, MS, Principal Investigator — University of Texas at Houston Medical School
Locations (1):
- University of Texas at Houston Medical School; Pediatric Nephrology and Hypertension Clinics, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Samuel JP, Samuels JA, Brooks LE, Bell CS, Pedroza C, Molony DA, Tyson JE. Comparative effectiveness of antihypertensive treatment for older children with primary hypertension: study protocol for a series of n-of-1 randomized trials. Trials. 2016 Jan 8;17:16. doi: 10.1186/s13063-015-1142-y. PMID 26746195
- [Derived] Samuel JP, Tyson JE, Green C, Bell CS, Pedroza C, Molony D, Samuels J. Treating Hypertension in Children With n-of-1 Trials. Pediatrics. 2019 Apr;143(4):e20181818. doi: 10.1542/peds.2018-1818. Epub 2019 Mar 6. PMID 30842257

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From June 2013 until July 2016, 55 patients were eligible based on inclusion/exclusion criteria, and 42/55 patients (76%) agreed to participate.
Pre-assignment Details: Forty-two children agreed to participate. Among the 30 patients taking antihypertensive medication prior to enrollment, 20 completed an updated baseline ambulatory BP monitoring. As a result, 23% (7/30) were found to be normotensive without medication, and did not undergo an n-of-1 trial. These 7 patients were not assigned to a treatment arm.
Period: First Intervention (2 Weeks)
Arm/Group | Amlodipine, Then HCTZ, Then Lisinopril | Amlodipine, Then Lisinopril, Then HCTZ | HCTZ, Then Amlodipine, Then Lisinopril | HCTZ, Then Lisinopril, Then Amlodipine | Lisinopril, Then Amlodipine, Then HCTZ | Lisinopril, Then HCTZ, Then Amlodipine
Started | 5 | 6 | 5 | 8 | 4 | 7
Completed | 5 | 5 | 4 | 8 | 4 | 6
Not Completed | 0 | 1 | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 0 | 1
Period: Second Intervention (2 Weeks)
Arm/Group | Amlodipine, Then HCTZ, Then Lisinopril | Amlodipine, Then Lisinopril, Then HCTZ | HCTZ, Then Amlodipine, Then Lisinopril | HCTZ, Then Lisinopril, Then Amlodipine | Lisinopril, Then Amlodipine, Then HCTZ | Lisinopril, Then HCTZ, Then Amlodipine
Started | 5 | 5 | 4 | 8 | 4 | 6
Completed | 5 | 5 | 4 | 8 | 4 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention (2 Weeks)
Arm/Group | Amlodipine, Then HCTZ, Then Lisinopril | Amlodipine, Then Lisinopril, Then HCTZ | HCTZ, Then Amlodipine, Then Lisinopril | HCTZ, Then Lisinopril, Then Amlodipine | Lisinopril, Then Amlodipine, Then HCTZ | Lisinopril, Then HCTZ, Then Amlodipine
Started | 5 | 5 | 4 | 8 | 4 | 6
Completed | 5 | 5 | 4 | 8 | 4 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects who participated in an n-of-1 trial received all three interventions in a cross-over fashion.
Groups:
- Participants Who Completed N-of-1 Trials: Participants who completed the first treatment cycle in the n-of-1 trial
Arm/Group | Participants Who Completed N-of-1 Trials
Number analyzed (Participants) | 32
Age, Continuous [Median (Full Range); unit: years] | 14 [9 to 19]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 20
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: The Number of Patients for Whom Each Drug is Selected as the Preferred Therapy
Description: For each n-of-1 trial, the preferred drug is defined as that which produces normal ambulatory blood pressure (by pediatric Ambulatory blood pressure monitoring (ABPM) standards), with the greatest magnitude of wake mean systolic BP reduction, and without unacceptable side effects.
Time Frame: The outcome of BP control and side effect tolerability will be assessed 2 weeks after starting each drug. Participants will be followed for an average of 10-12 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Lisinopril | Amlodipine | Hydrochlorothiazide
Number analyzed (Participants) | 32 | 32 | 32
Participants | 16 | 8 | 4

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Lisinopril | Amlodipine | Hydrochlorothiazide
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 0/32 | 0/32 | 2/32
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lisinopril (N=32) | Amlodipine (N=32) | Hydrochlorothiazide (N=32)
Hypokalemia (Investigations) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes